CLINICAL TRIAL: NCT06382012
Title: Antiemetic Fosaprepitant To Remedy Nausea and Vomiting
Acronym: AFTR NV RCT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-15703
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Nausea and Vomiting; Nausea; Vomiting
Keywords: Fosaprepitant; Nausea and Vomiting; Nausea; Vomiting; Randomized Control Trial; Ondansetron; Adults
MeSH Terms: conditions — Nausea; Vomiting | interventions — fosaprepitant; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Intervention (Experimental): Fosaprepitant 150mg IV administered over 15 minutes
  Interventions: Drug: Fosaprepitant 150 mg
- Standard-of-Care Intervention (Active Comparator): Ondansetron 4mg IV administered over 15 minutes
  Interventions: Drug: Ondansetron 4 mg

INTERVENTIONS:
Drug: Fosaprepitant 150 mg — Fosaprepitant 150mg IV administered over 15 minutes
  Arms: Investigational Intervention
Drug: Ondansetron 4 mg — Ondansetron 4mg IV administered over 15 minutes
  Arms: Standard-of-Care Intervention

SUMMARY:
The study team proposes a randomized, double-blind, RCT to address the following goal: to determine the relative efficacy and adverse event profile of fosaprepitant compared to the standard of care antiemetic ondansetron. Fosaprepitant and its active metabolite aprepitant are a relatively new class of antiemetic that exclusively acts in the central nervous system by blocking neurokinin (NK-1) which is a key signaling molecule in the centrally mediated aspects of the vomiting reflex. Currently, fosaprepitant and aprepitant both have only two United Stated Food and Drug Administration (USFDA) approved indications for nausea and vomiting: chemotherapy-induced and postoperative. Neurokinin inhibitors are highly effective and generally well-tolerated. Therefore, this class of medication may be a more appropriate medication for the millions of patients with nausea and vomiting that seek care in EDs. Intravenous fosaprepitant is converted to the active metabolite aprepitant on the order of minutes and is significantly cheaper to procure at this time. The outcome for the efficacy analysis will be no need for additional medication to treat nausea and vomiting within 2 hours of investigational medication administration. The primary outcome for the tolerability analysis will be the development of any new symptom within 2 hours of medication administration.

DETAILED DESCRIPTION:
Nausea and vomiting (NV) are common and interrelated conditions. Approximately 50% of adults experience nausea in a given year while 30% of adults experience vomiting over the same period. Of this population of symptomatic individuals with NV, 25% of patients seek care in any healthcare delivery setting. Health Care Utilization Project (HCUP) data indicates that nearly 9.0 million patients seek care for NV in emergency departments (EDs) each year in the United States.

Antiemetics are used to treat NV. Antiemetics currently utilized in the emergency department setting for NV do not always work on the first dose and have a plethora of side effects because of their peripheral mechanism of action outside of the vomiting reflex pathway in the central nervous system. These medications include ondansetron, promethazine, metoclopramide, olanzapine, haloperidol. Chief among these side effects is alteration of an aspect cardiac electrical signaling called the QT segment which represents the duration of ventricular contraction and relaxation. The QT segment is prolonged with commonly used antiemetics which can often be a prelude to cardiac dysrhythmias that are associated with mortality. As a result, patients with NV often have long length-of-stay (LOS) involving supportive care with intravenous fluids or empiric treatment with medications that can potentiate development of cardiac dysrhythmias. This is a problem in busy emergency departments (EDs) struggling to accelerate patient throughput in order to appropriately keep up with patient volume in an under-supplied hospital bed environment nationally.

Fosaprepitant and its active metabolite aprepitant are a relatively new class of antiemetic that exclusively acts in the central nervous system by blocking neurokinin (NK-1) which is a key signaling molecule in the centrally mediated aspects of the vomiting reflex. Currently, fosaprepitant and aprepitant both have only two United Stated Food and Drug Administration (USFDA) approved indications for nausea and vomiting: chemotherapy-induced and postoperative. Neurokinin inhibitors are highly effective and generally well-tolerated. Therefore, this class of medication may be a more appropriate medication for the millions of patients with nausea and vomiting that seek care in EDs. Intravenous fosaprepitant is converted to the active metabolite aprepitant on the order of minutes and is significantly cheaper to procure at this time.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old
* Present to an emergency department (ED) for nausea and/or vomiting as defined by the International Classification of Diseases (ICD-10), or identified by treating clinician
* Following the approval of a protocol amendment, study patients who have received an antiemetic and remain persistently nauseated after 2 hours will be eligible to participate in the study

Exclusion Criteria:

* Pregnancy, desiring pregnancy, or lactating
* Antiemetic medication use less than 2 hours prior to screening
* Bradycardia (heart rate less than 60 bpm heart rate)
* Prolonged QTc (>480ms)
* Not conversant in English or Spanish
* Altered mental status
* Dementia
* Lack of phone for follow-up communication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sustained Relief from NV | 24 hours (measured every 15 minutes for the first 2 hours, then hourly after that until disposition; reassessed at 24 hours)
  Sustained relief from nausea and vomiting will be determined by the intensity of nausea reported by participants following administration of antiemetic. Intensity of nausea will be reported as either None, Mild, Moderate, or Severe. The number/percentage of participants reporting each degree of nausea intensity will be summarized
  Sustained relief of nausea and vomiting requires a patient to present with a nausea intensity of either "severe" or "moderate," which is then reduced by treatment to at least "mild" or "none," within two hours of medication administration, and then maintained at "mild" or "none" level for the entire 24-hour period following medication administration without the use of rescue medication.

SECONDARY OUTCOMES:
Severity of Nausea | 24 hours (measured every 15 minutes for the first 2 hours, then hourly after that until disposition; reassessed at 24 hours)
  Mean severity of nausea scores will be evaluated and summarized based on a visual analogue scale from 0 to 100 (0 = no nausea, 100 = worst nausea possible)
Need for rescue antiemetic medication | 2 hours (assessed at the 2 hour mark after administration of the intervention)
  Binary outcome for needing or not needing additional dosing of antiemetic medication to treat nausea will be determined
Medication Preference | 24 hours
  Participant preference for receiving the same antiemetic medication as administered for a subsequent episode of nausea and vomiting will be determined. Binary (Yes/No) responses will be summarized
Functional disability | 24 hours (assessed prior to receiving intervention, at 2 hour point after receiving intervention, and 24 hours after intervention)
  Patient reported functional disability will be assessed. Functional disability will be categorized as either severe, moderate, mild, or not impaired, and summarized
Vomiting | 24 hours
  The mean number of vomiting episodes per patient will be assessed and summarized
Hospitalization | 24 hours
  The percentage of patients who require hospitalization within 24 hours due to NV symptoms will be determined
Fluid Treatment | 4 hours
  The percentage of patients treated with IV fluids will be determined
Mean Fluid Volume | 4 hours
  The mean per patient volume of IV fluids administered will be summarized
Length of Stay | Initial presentation to disposition, approximately 4 hours
  Mean length of stay, defined as the interval of time from initial presentation to disposition, will be determined
QTc Interval (QT interval corrected for heart rate) | Prior to Intervention and at disposition, approximately 2 hours
  Mean QTc durations, as calculated from ECG readings administered prior to receiving intervention and at disposition, will be determined. Prolonged QT interval is commonly associated with antiemetics and can often be a prelude to cardiac dysrhythmias associated with mortality
Revisit Rate | 24 hours
  Revisit rate will be assessed as the number/percentage of participants requiring a revisit to the Emergency department for NV

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center (Montefiore and Weiler EDs), The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mechanisms and Control of Emesis: A Satellite Symposium of the European Neuroscience Association: Proceedings of an International Meeting Held in Marseille (France), 4-7 September 1992. John Libbey Eurotext
- [Background] Singh P, Yoon SS, Kuo B. Nausea: a review of pathophysiology and therapeutics. Therap Adv Gastroenterol. 2016 Jan;9(1):98-112. doi: 10.1177/1756283X15618131. PMID 26770271
- [Background] Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Available from http://www.ncbi.nlm.nih.gov/books/NBK52651/ PMID 21413206
- [Background] Pourmand A, Mazer-Amirshahi M, Chistov S, Sabha Y, Vukomanovic D, Almulhim M. Emergency department approach to QTc prolongation. Am J Emerg Med. 2017 Dec;35(12):1928-1933. doi: 10.1016/j.ajem.2017.08.044. Epub 2017 Aug 24. PMID 28855066
- [Background] Franklin BJ, Vakili S, Huckman RS, Hosein S, Falk N, Cheng K, Murray M, Harris S, Morris CA, Goralnick E. The Inpatient Discharge Lounge as a Potential Mechanism to Mitigate Emergency Department Boarding and Crowding. Ann Emerg Med. 2020 Jun;75(6):704-714. doi: 10.1016/j.annemergmed.2019.12.002. Epub 2020 Jan 23. PMID 31983501
- [Background] Aapro M, Carides A, Rapoport BL, Schmoll HJ, Zhang L, Warr D. Aprepitant and fosaprepitant: a 10-year review of efficacy and safety. Oncologist. 2015 Apr;20(4):450-8. doi: 10.1634/theoncologist.2014-0229. Epub 2015 Mar 20. PMID 25795636
- [Background] Langford P, Chrisp P. Fosaprepitant and aprepitant: an update of the evidence for their place in the prevention of chemotherapy-induced nausea and vomiting. Core Evid. 2010 Oct 21;5:77-90. doi: 10.2147/ce.s6012. PMID 21042544
- [Background] Furyk JS, Meek RA, Egerton-Warburton D. Drugs for the treatment of nausea and vomiting in adults in the emergency department setting. Cochrane Database Syst Rev. 2015 Sep 28;2015(9):CD010106. doi: 10.1002/14651858.CD010106.pub2. PMID 26411330
- [Background] Yang Y, Yang N, Wu L, Ouyang Q, Fang J, Li J, Liao W, Cai K, Huang J, Li J, Zhang Y, Wang X, Zhang H, Xu N, Zhao Q, Hu X, Li W, Zhong W, Zhong D, Cheng G, Ye S, Zhong M, Wang D, Liu H, Zheng J, Liu X, Xu H, Zhang L. Safety and efficacy of aprepitant as mono and combination therapy for the prevention of emetogenic chemotherapy-induced nausea and vomiting: post-marketing surveillance in China. Chin Clin Oncol. 2020 Oct;9(5):68. doi: 10.21037/cco-20-160. PMID 33161724
- [Background] Tramer MR, Phillips C, Reynolds DJ, McQuay HJ, Moore RA. Cost-effectiveness of ondansetron for postoperative nausea and vomiting. Anaesthesia. 1999 Mar;54(3):226-34. doi: 10.1046/j.1365-2044.1999.00704.x. PMID 10364857